CLINICAL TRIAL: NCT03524547
Title: Comparison of Endotracheal Tube Shapes for Intubation With Videolaryngoscope in Normal Airways
Brief Title: Endotracheal Tube Shapes for Intubation With Videolaryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-01-033-001; 2018-01-016-003 (Other: Hanyang university hospital)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- J-shaped (Experimental): Endotracheal tube will be molded into a J-shape that is similar to that of Macintosh type blade of a McGrath MAC® videolaryngoscope.
  Interventions: Device: J shaped stylet used for endotracheal intubation
- 60-degrees (Active Comparator): Endotracheal tube will be bent 60 degrees.
  Interventions: Device: 60-degrees stylet used for endotracheal intubation

INTERVENTIONS:
Device: J shaped stylet used for endotracheal intubation — After inserting a stylet into the endotracheal tube, the tube will be molded into a J-shape.
  Arms: J-shaped
Device: 60-degrees stylet used for endotracheal intubation — After inserting a stylet into the endotracheal tube, the tube will be bent 60-degrees.
  Arms: 60-degrees

SUMMARY:
In this study, investigators will compare the efficacy of two shapes of endotracheal tube molded by stylet in endotracheal intubation using videolaryngoscope (McGrath MAC®). The participants will randomly be divided into two groups; J-shaped tube and 60-degrees-curved tube.

DETAILED DESCRIPTION:
Since the intubation using videolaryngoscope does not need straightened oral-pharyngeal-laryngeal axis, certain curvature of endotracheal tube is needed for the successful intubation using the videolaryngoscope.

Participants in both groups will be intubated with videolaryngoscope (McGrath MAC®). Stylet will be inserted in the endotracheal tubes and will be bent to a specific shape by the assigned group. In the J-shaped tube group, endotracheal tube will be molded to a shape similar to the blade of the videolaryngoscope (McGrath MAC®). In the 60-degrees-curved tube group, endotracheal tube will be bent 60 degrees. Time to intubation, intubation attempts and ease of intubation wil be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for the surgery under general anesthesia
* Adult patients from 18 years to 65 years
* American society of Anesthesiologist physical status 1,2,3

Exclusion Criteria:

* Previously diagnosed for the difficult intubation
* Pregnancy
* Obesity (Body mass index over 40 g/m^2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Time to intubate | 20 minutes after induction started.
  the time took from the blade passing through the incisor teeth of the patient to the first end tidal CO2 appears on the anesthesia monitor screen.

SECONDARY OUTCOMES:
Numbers of intubation attempts | 20 minutes after induction started.
  numbers of attempts for the successful endotracheal intubation
Level of difficulty in intubation | 20 minutes after induction started.
  easy, moderate, difficult

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, M.D., Principal Investigator — Kangbuk Samsung Hospital; Hyunyoung Lim, M.D., Principal Investigator — Hanyang University
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided